CLINICAL TRIAL: NCT03694691
Title: Development of a Liver Viability Index for Transplantation
Brief Title: Developing Viability Index for Machine Perfused Livers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Heidi Yeh, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Liver Perfusion ATP
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy (Experimental): Biopsies taken at protocol specified time points
  Interventions: Diagnostic Test: Liver Biopsy

INTERVENTIONS:
Diagnostic Test: Liver Biopsy — For measurement of tissue co-factor levels, we will take needle biopsies of transplanted livers immediately after procurement, immediately prior to implantation (at the end of preservation), 30 minutes after portal vein reperfusion, and 30 minutes after hepatic artery reperfusion. For those livers that have more than 60 minutes between portal vein and hepatic artery reperfusion, an additional biopsy will be performed at 60 minutes after portal vein reperfusion. Post-procurement biopsies will be collected regardless of where the liver was obtained.

SUMMARY:
Machine perfusion technology is nearing the point of rescuing discarded liver grafts in the hope of proving them to be or improving them to the point of being transplantable. However, there are no validated metrics to determine transplantability after machine perfusion. This study involves collecting biopsies from transplanted livers before and after implantation to correlate metabolite and gene expression with post-transplant function. This data will help develop a viability index for machine perfused livers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-75 years of age.
* Candidate for a deceased-donor liver allograft.

Exclusion Criteria:

* Seropositivity for HIV-1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak transaminase value post transplant | 1 Year
  The primary endpoint is peak transaminase values since transaminase elevation is a marker of hepatocyte injury

SECONDARY OUTCOMES:
Acute Liver Rejection | 1 Year
Incidence of major Infection | 1 Year
Hepatitis C Recurrence (in Hepatitis C positive recipients) | 1 Year
Kidney Failure | 1 Year
Biliary Complications | 1 Year
Liver Graft Failure | 1 Year
Death | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Yeh, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No